CLINICAL TRIAL: NCT01551238
Title: Energy Expenditure and Sleep in Response to Protein/Carbohydrate and Fat Ratio
Brief Title: Energy Expenditure, Sleep and Macronutrients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL39152
Record Dates: First submitted 2011-12-14; First posted 2012-03-12 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Overweight; Overnutrition; Nutrition Disorders; Body Weight; Signs and Symptoms
Keywords: Energy expenditure; Sleep; Protein; Carbohydrate
MeSH Terms: conditions — Obesity; Overweight; Overnutrition; Nutrition Disorders; Body Weight; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein intake of 5 energy percent (Experimental)
  Interventions: Dietary Supplement: Differences in protein content of meals
- Protein intake of 30 energy percent (Experimental)
  Interventions: Dietary Supplement: Differences in protein content of meals

INTERVENTIONS:
Dietary Supplement: Differences in protein content of meals — Differences in protein content (energy percent) of meals
  Arms: Protein intake of 5 energy percent
Dietary Supplement: Differences in protein content of meals — Differences in protein content (energy percent) of meals
  Arms: Protein intake of 30 energy percent

SUMMARY:
The purpose of this study is to determine energy expenditure and sleep in response to protein/carbohydrate and fat ratio of the diet over a short-term and long-term period of time.

DETAILED DESCRIPTION:
The prevalence of obesity has increased worldwide to epidemic proportions. For long-term treatment success permanent lifestyle changes are necessary with regard to approach to food, physical activity patterns and behavior to emotional stress. Moreover, an association has been shown between sleep disturbance and obesity. Weight loss strategies regarding food intake regulation mainly focused on changing patterns of fat and carbohydrate consumption during the last decades. The role of protein has largely been ignored. However, protein has been observed to increase satiety and energy expenditure to a greater extent than carbohydrate and fat and can therefore reduce energy intake. However, it still has to be confirmed if this effect is permanent or transient over a longer period of time. Moreover, dietary intakes may significantly affect sleep when macronutrient intakes are manipulated. Since sleep deprivation has been recognized as a risk factor for obesity, improving sleep by a change in macronutrient intake would be promising in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age between 18-35 years
* BMI 18-27 kg/m2
* non-smoking
* weight stable (weight change < 3 kg during the last 6 months)
* no sleeping problems
* not using a more than moderate amount of alcohol (> 10 consumptions/wk)
* not using medication or supplements except for oral contraceptives in women

Exclusion Criteria:

* not healthy
* do not meet the criteria for BMI and age
* smoking
* not being weight stable
* using medication or supplements except for oral contraceptives in women
* sleeping problems
* using a more than moderate alcohol consumption
* pregnant or lactating
* allergic for the used food items

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
energy expenditure | 48 hours
substrate oxidation | 48 hours
sleep | 48 hours

SECONDARY OUTCOMES:
body composition | 48 hours
fat distribution | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Margriet S. Westerterp-Plantenga, Prof. dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Department of Human Biology, Nutrition and Toxicology Research Institute Maastricht (NUTRIM), Maastricht, Netherlands

REFERENCES:
- [Derived] Hursel R, Martens EA, Gonnissen HK, Hamer HM, Senden JM, van Loon LJ, Westerterp-Plantenga MS. Prolonged Adaptation to a Low or High Protein Diet Does Not Modulate Basal Muscle Protein Synthesis Rates - A Substudy. PLoS One. 2015 Sep 14;10(9):e0137183. doi: 10.1371/journal.pone.0137183. eCollection 2015. PMID 26367529
- [Derived] Martens EA, Gonnissen HK, Gatta-Cherifi B, Janssens PL, Westerterp-Plantenga MS. Maintenance of energy expenditure on high-protein vs. high-carbohydrate diets at a constant body weight may prevent a positive energy balance. Clin Nutr. 2015 Oct;34(5):968-75. doi: 10.1016/j.clnu.2014.10.007. Epub 2014 Nov 8. PMID 25466951
- [Derived] Martens EA, Gatta-Cherifi B, Gonnissen HK, Westerterp-Plantenga MS. The potential of a high protein-low carbohydrate diet to preserve intrahepatic triglyceride content in healthy humans. PLoS One. 2014 Oct 16;9(10):e109617. doi: 10.1371/journal.pone.0109617. eCollection 2014. PMID 25330327